CLINICAL TRIAL: NCT02884427
Title: Effects of Ascending and Descending Direct Current on Grip Strength. Evaluation Through Dynamometry and Myofeedback. Randomized, Controlled Trial.
Brief Title: Direct Current Cathode and Anode Effects and Changes in Handgrip Strength. Evaluation Through a Dynamometer Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 60312061
Record Dates: First submitted 2016-08-15; First posted 2016-08-31 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Handgrip Strength
Keywords: Direct current; Dynamometry; Hand strength; Electrotherapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cathode Stimulation (Experimental): Group that is involved with the (black) negative electrode seeking the polar effect of nervous increased excitability and conductivity with the current application.
  Interventions: Device: Cathode stimulation
- Anode Stimulation (Experimental): Group that is involved with the (red) positive electrode seeking the polar effect of nervous excitability and conductivity decreased with the current application.
  Interventions: Device: Anode stimulation
- Control (Placebo Comparator): Group that will be placed electrotherapy without operation, but only installation. Patients in this group will see the team work but it will not be delivering current.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Cathode stimulation — Electrical stimulation through the cathode or negative pole, in which a peripheral nerve will be subject to the passage of a direct current seeking increased excitability and conductivity during the passage of current.
  Other Names: Cathode Polar effect
  Arms: Cathode Stimulation
Device: Anode stimulation — Electrical stimulation through the anode or positive pole, in which a peripheral rib will be subjected to the passage of a direct current seeking to reduce excitability and conductivity during the passage of current.
  Other Names: Anode Polar effect
  Arms: Anode Stimulation
Device: Placebo — Current application without the actual electric conduction to the person occurs. This will be achieved by adjusting parameters while installing another channel and not one that is working.
  Other Names: Non intervention
  Arms: Control

SUMMARY:
The design aims to investigate the value of direct current, specifically the polar effects this has, and its influence on neuromuscular changes described in the literature. This research proposal seeks to assess the influence of application anode and cathode pole in muscle strength when testing handgrip dynamometry by healthy subjects. The study will evaluate changes in muscle strength when performing a manual dynamometer test in a group exposed to the application of cathode, another exposed to the application of anode, compared with a control that will not receive the intervention will be evaluated. Subsequently the investigators proceed to compare the maximum force obtained from the dynamometry test in each of groups and between the groups .

DETAILED DESCRIPTION:
1. Methodology

This research has the characteristics of a random analytical experimental design (ECA). The study was conducted in the laboratory of physiotherapy, room 401, 4th floor, building C5 University Andres Bello (UNAB), Faculty of Rehabilitation Sciences, Campus Casona, Nº700 Street Fernández Concha, Santiago, Chile. The sample was selected from the university population that is part of the faculty. The study was submitted to the ethics committee of the East Metropolitan Health Service (SSMO) of Salvador Hospital. Once approved by the ethics committee began the investigation. It was taken as population all students of the Faculty of Rehabilitation Sciences, made up of races Physical Therapy, Speech Therapy and Occupational Therapy. The study group was determined through a simple random sampling process, which was conducted through a questionnaire with closed questions. This questionnaire allowed select participants according to the inclusion and exclusion criteria proposed in the work. The number of participants was taken for the convenience of researchers. The final sample included 150 participants. Student population share similar characteristics, so that most made them compatible for the sample. Inclusion criteria were established: participants aged 18 years and people that they should not discomfort or pain on the handgrip. Moreover Exclusion criteria were considered: muscle pathologies skeletal hand, wrist or elbow in the last 6 months, the presence of materials osteosynthesis or endoprosthesis in areas of application, peripheral neurological diseases such as neuropraxias or nervous cuts, skin disorders application areas, such as burns, wounds, scars, apprehension or fear of the application of electrotherapy, non-completion of the evaluation protocol / intervention designed for studio or away from it, and do not sign the consent for participation.

3 stages of conducting the study were designated. Stage 1 called "The Sample Phase", had a duration of one week. This Phase consisted of the implementation of the survey to students, followed by analysis of the collected information and registration for a first filter potential participants. The survey was applied to all courses of the Faculty of Rehabilitation Sciences. The first filter was given with the survey questions that has specifics questions with the inclusion and exclusion criteria. Participants who met the characteristics of participation and were invited to join the study. The students will be contacted personally. Students interested will be explained in detail the study and were asked to give their written consent. Informed consent reflected the 4 principles of bioethics so as to safeguard the integrity of each person.

The second stage of design called "Evaluation Phase" lasted 5 days. In this phase the ability to perform hand grip on the participants according to the protocol established in the investigation was assessed. The strength assessment will be probe in the same conditions in which they worked on the study. At this level, people explained everything concerning the characteristics of electrical stimulation used, and as applicable. This stage marked a second filter instance dismissing students who had discomfort or inability to perform the handgrip. After this phase had the final number of participants who made up the final sample of the study, giving way to step 3.

The stage called "Experimentation Phase" had a duration of 3 weeks. The sample was randomly so as to establish three working groups, a group called "Cathode Stimulation", another group called "Anode Stimulation" and a third group called "Control Group". The group "Cathode stimulation" includes 48 participants, while the "Anode Group" had 52 participants and the "Group Control" 50 participants.

The designation of each group participants, was conducted by the director of the study, by simple randomization process, through Microsoft Excel® program. This allowed decrease selection bias. After this process the director conduce each student to the box in which the force will be evaluated. A first evaluator (Evaluator 1) analyzed the demographic characteristics of each group, including age, body mass index (BMI), and gender, which allowed determine the characteristics per group. This would establish any comparisons at the end of work, taking the results. This information is obtained by the survey. The participants of the 3 groups were evaluated by another evaluator (Evaluator 2), who recorded the average maximum handgrip force developed by the dominant limb of the participants. Grip strength was evaluated according to the evaluation protocol proposed by manual torque test, registering kilograms (kg) of force developed by understanding. The evaluation included 3 executions leaving a rest interval of 15 seconds between each attempt (measurement protocol). The evaluator 2 recorded in an Excel spreadsheet the initial 3 attempts, leaving the best maximal force value of them as definitive. This was considered as the maximal handgrip Force value prior the intervention. After the director derived each participant according to the particulary group, Cathode, Anode or Control. The design featured participation of three therapists, one for each working group.

Therapist did not know the data obtained from the evaluation of strength, and the students that belonged the groups. Physiotherapists executors were familiar with the application of electric current. Each therapist worked using direct current with 500 COMBI GYMNA® equipment company. In the application we worked with one channel team, applying an electrode on the engine of the flexor muscles of the forearm dominant point and the other electrode closing the circuit on the side face of the opposite arm. It was taken as described by the motor point SENIAM corporation, who recommend specific motor points for the application surface electromyography. For the Cathode group the black electrode was used in the forearm muscle flexor of the dominant side for the anode group red electrode was used in the forearm muscle flexor of the dominant side, while for the control group the black electrode was used in the same musculature. The first two groups were given a current intensity of 2mA (based on the safety recommendations when applying direct current), while the control group was not applied current. With these parameters a current density of 0,04mA /cm2 was obtained. (rubber electrodes coal rectangular area 48cm2). Each therapist was masked output color channel electrode by a black tape, so that it was not known what was the black or red electrode. The treatment time for each group was 10 minutes, according to the protocol established for the investigation. This generated a dose of current 5mA/min. Participants of the three groups were installed on wooden stretchers sitting in Fowlers position maintaining a 45 ° angle. The electrode was placed on the side of the dominant limb with the device screen facing towards the foot of the participant, so the person could not display the current value set. After the application of the current, the participants left the room intervention and were led by the director to the force assessment room. In this room would register the best post maximum grip strength. The evaluator recorded three attempts, leaving the same time of 15 seconds between each. The evaluator 1 record average of the 3 values in an Excel spreadsheet. This is the value designated as post test (maximal strength post intervention).

After completing the measurements two weeks were available to sort the data and the analysis of the recorded information. This task was driven by the research director who was responsible for storing and sorting data received by the evaluators. The Microsoft Excel program was used for this process register all data. Descriptive statistics for the maximum strength was represented in the form of averages, frequencies and standard deviation. This information is also represented as graphs of boxes comparing IMC, gender and age per group. Inferential statistics was development with the Shapiro Will test to determinate a normally distributed data, then using ANOVA test or T-test. For data not normally distributed Kruskal-Wallis test was applied. The statistics was perform with de STATA program. Once the statistical analysis done within 3 weeks for the analysis of results, and approach the discussion and results are considered.

2. Measurement handgrip strength protocol pre and post electrotherapy

Measuring handgrip strength will be conducted in the laboratory of physiotherapy, room 401, 4th floor, building C5 University Andres Bello (UNAB), Faculty of Rehabilitation Sciences, Campus Casona, Las Condes, Street Fernández Concha Nº700, Santiago, Chile. Initially, participants were instructed to sit in a straight chair with dimensions of 42cm high, 46 cm wide by 40 cm long, back tilt of 10 ° and dimensions of 43 cm high by 46 cm wide, the participant shall be placed with his feet flat on the floor, erect trunk in contact with the back, head and neck in a neutral position, shoulder adducted, in neutral rotation, elbow bent at 90, forearm prone neutral supination, unsupported any surface and wrist position neutra.67 for the test, a hydraulic hand dynamometer model Dynatron® which has a weight of 600g, dimensions of 26 cm long by 13 cm wide, with reading will be used dual measurement scale up to 200lbs / 90kg, also has five levels of manual adjustment, which will be set at the second level. The estimated time measuring participant is 2 minutes.

The handgrip strength was measured on 3 occasions, the break between measurements is 15 seconds, taking an estimated 54 seconds net force measurement by participant time. Participants will be instructed to position themselves correctly in the workstation and apply maximum force for 3 seconds and work at maximum effort in each test returning the marker measuring instrument 0 lbs / after each measurement kg. The evaluator register the average maximal handgrip strength between the 3 attempts. For the data registration we will use Microsoft Excel® program. The division consist in 3 categories of participants, Cathode Group, Anode Group and Control Group. The pre electrotherapy application data will be recorded immediately after the measurement of palmar force dynamometry.

2. Electrotherapy Protocol

The intervention will take place in the laboratory of physiotherapy, room 401, 4th floor, building C5 University Andres Bello (UNAB), Faculty of Rehabilitation Sciences, Campus Casona, Las Condes, Street Fernández Concha Nº700, Santiago , Chile. After the initial force measurement participants will be placed in the particular station for applying electrotherapy, where each participant will be instructed to position themselves in a sitting position 45º on a stretcher fixed two bodies, with dimensions 190cm long by 70cm wide and 80cm high, each participant must support the trunk on the top of the table, inclined at 45 degrees, with both elbows, forearms and arms bare skin, well supported on the stretcher.

For the application of electrotherapy was applied with the devise Gymna® Combi 500 model, which it is characterized by having a unit of electrotherapy, ultrasound and laser.

It was also be used carbon electrodes which measurements are 7.5cm long x 6cm wide with their respective terminals, 2 driving pads 9.5 cm long by 8 cm wide and 2 fasteners with velcro for electrodes, 47cm long by 5 cm wide.

During the intervention, it proceeds to plug the equipment into an outlet 220v conventional power, then connect the electrodes in one of the two channels available on the device. Once the participant is correctly positioned in the workstation, the therapist will place correctly the electrodes, applying an electrode on the belly of the flexor muscles of the forearm (established on the recommendation of SENIAM project point), and the other electrode closing the circuit laterally on the other forearm. For the Cathode Group the black electrode is used in the flexor muscles of the dominant hand, for the Anode Group red electrode is used in the flexor muscles of the dominant hand, while the Control Group the black electrode will be used in the same muscles, procedure will be repeated for the 3 groups of participants, once completed this procedure. The Therapist applied to the first two groups a current of 2mA, thereby determining a density 0,04mA current /cm2 considering a size of 48cm2 electrode, while the control group will not be applied any intensity keeping the power on but without emission. For the 3 groups of participants application time is 10 electrotherapy minutes.

ELIGIBILITY:
Inclusion Criteria:

* Participants older than 18 years
* Do not manifest discomfort or pain when performing the handgrip.

Exclusion Criteria:

* Skeletal muscle pathologies in hand, wrist or elbow in the last 6 months.
* Materials osteosynthesis or endoprosthesis in areas of application.
* Peripheral neurological pathologies as neuropraxias or nerve sections.
* Changes in the skin of the application areas, such as burns, wounds, scars.
* Apprehension or fear of the application of electrotherapy.
* No completion of the evaluation protocol / intervention, designed for study or abandonment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hernán Andrés HB de la Barra Ortiz, Mg., Principal Investigator — University Teacher and Physical therapist
Locations (1):
- Universidad Andrés Bello, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michelle H. Cameron, Physical Agents in Rehabilitations 2003, Elsevier. Cap. VIII, P, 220.
- [Background] Currier DP, Mann R. Muscular strength development by electrical stimulation in healthy individuals. Phys Ther. 1983 Jun;63(6):915-21. doi: 10.1093/ptj/63.6.915. PMID 6856678
- [Background] Thurin E, Meehan PF, Gilbert BS. Treatment of pain by transcutaneous electric nerve stimulation in general practice. Med J Aust. 1980 Jan 26;1(2):70-1. doi: 10.5694/j.1326-5377.1980.tb134629.x. PMID 6965758
- [Background] Rodríguez Martin JM, Corrientes más utilizadas en la Electroterapia en Fisioterapia. Editorial Medica Panamericana, Cap II, P. 61- 86, 2000.
- [Background] Glass JM, Stephen RL, Jacobson SC. The quantity and distribution of radiolabeled dexamethasone delivered to tissue by iontophoresis. Int J Dermatol. 1980 Nov;19(9):519-25. doi: 10.1111/j.1365-4362.1980.tb00380.x. PMID 7429701
- [Background] Conjeevaram R, Banga AK, Zhang L. Electrically modulated transdermal delivery of fentanyl. Pharm Res. 2002 Apr;19(4):440-4. doi: 10.1023/a:1015135426838. PMID 12033377
- [Background] Petelenz TJ, Buttke C, Bonds LB, Lloyd JE, Beck RL, Stephens SC. Iontophoresis of dexamethasone: laboratory studies. J Controll Rel 1992;20:55-66.
- [Background] Fujita M, Hukuda S, Doida Y. The effect of constant direct electrical current on intrinsic healing in the flexor tendon in vitro. An ultrastructural study of differing attitudes in epitenon cells and tenocytes. J Hand Surg Br. 1992 Feb;17(1):94-8. doi: 10.1016/0266-7681(92)90021-s. PMID 1640154
- [Background] Raiman J, Koljonen M, Huikko K, Kostiainen R, Hirvonen J. Delivery and stability of LHRH and Nafarelin in human skin: the effect of constant/pulsed iontophoresis. Eur J Pharm Sci. 2004 Feb;21(2-3):371-7. doi: 10.1016/j.ejps.2003.11.003. PMID 14757511
- [Background] Kalia YN, Naik A, Garrison J, Guy RH. Iontophoretic drug delivery. Adv Drug Deliv Rev. 2004 Mar 27;56(5):619-58. doi: 10.1016/j.addr.2003.10.026. PMID 15019750
- [Background] Panus PC, Ferslew KE, Tober-Meyer B, Kao RL. Ketoprofen tissue permeation in swine following cathodic iontophoresis. Phys Ther. 1999 Jan;79(1):40-9. PMID 9920190
- [Background] Meijinde Faide R. Rodriguez .Villamil Fernandez JLy Teiro Vidal J. Corrientes Galvanicas En. Martinez Morillo M, Pastor Vega, y Sandra Portero F. Manual de Medicina Fisica Harcourt Brace España 1998 P150-68.
- [Background] Kvandal P, Stefanovska A, Veber M, Kvernmo HD, Kirkeboen KA. Regulation of human cutaneous circulation evaluated by laser Doppler flowmetry, iontophoresis, and spectral analysis: importance of nitric oxide and prostaglandines. Microvasc Res. 2003 May;65(3):160-71. doi: 10.1016/s0026-2862(03)00006-2. PMID 12711257
- [Background] Guy RH, Delgado-Charro MB, Kalia YN. Iontophoretic transport across the skin. Skin Pharmacol Appl Skin Physiol. 2001;14 Suppl 1:35-40. doi: 10.1159/000056388. PMID 11509905
- [Background] Calvo Arenilla JI, Rubio López I. Iontoforesis. Aplicaciones de la Iontoforesis. Electroestimulaciónaplicada. En: Meaños Melón E, Alonso Martínez M, Murga Rodríguez F, Pinsach Ametller J, et al. Vigo: Obradoiro Gráfico; 2003. p. 157-172.
- [Background] Kahn J. Iontophoresis. Phys Ther. 1984 Jun;64(6):956, 959. doi: 10.1093/ptj/64.6.956a. No abstract available. PMID 6728918
- [Background] Oh SY, Guy RH. Effects of iontophoresis on electrical properties of human skin in vivo. Int J Pharmacol 1995;124:137-42.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cathode Stimulation | Anode Stimulation | Control
Started | 48 | 52 | 50
Completed | 48 | 52 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cathode Stimulation | Anode Stimulation | Control | Total
Number analyzed (Participants) | 48 | 52 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 11 | 24
  Between 18 and 65 years | 41 | 46 | 39 | 126
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (3) | 23 (2) | 22 (3) | 23 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 24 | 63
  Male | 30 | 31 | 26 | 87
Region of Enrollment [Number; unit: participants]
  Chile | 48 | 52 | 50 | 150
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24 (3) | 24 (3) | 25 (5) | 24 (3)

OUTCOME MEASURES:

1. Primary Outcome: Difference of Maximum Grip Strength
Description: The difference in maximum grip strength is that value in kilograms obtained between the best score of the first three gripping attempts made before the intervention compared to the best result obtained from the three attempts after the intervention. The maximum force difference will express the force changes before and after the participants are exposed to one of the treatments.
Time Frame: Baseline and 1 hours later (1 session of treatment), assessed as up to 1 month.
Measure: Mean (Standard Deviation); unit: Kilograms (Kg)
Arm/Group | Cathode Stimulation | Anode Stimulation | Control
Number analyzed (Participants) | 48 | 52 | 50
Kilograms (Kg) | 03 (5) | 0 (4) | -02 (5)

2. Secondary Outcome: Difference of Maximum Grip Strength for Males
Description: The difference in maximum grip strength for males is that value in kilograms obtained between the best score of the first three gripping attempts made before the intervention compared to the best result obtained from the three attempts after the intervention considering only the men of each group. Maximum force difference will express the force changes before and after the participants are exposed to one of the treatments.
Time Frame: Baseline and 1 hours later (1 session of treatment), assessed as up to 1 month.
Measure: Median (Inter-Quartile Range); unit: Kilograms (Kg)
Arm/Group | Cathode Stimulation | Anode Stimulation | Control
Number analyzed (Participants) | 30 | 31 | 26
Kilograms (Kg) | 1 [-3 to 4] | 0 [0 to 2] | 0.5 [-2 to 2]

3. Secondary Outcome: Difference of Maximum Grip Strength for Females
Description: The difference in maximum grip strength for females is that value in kilograms obtained between the best score of the first three gripping attempts made before the intervention compared to the best result obtained from the three attempts after the intervention considering only the women of each group. Maximum force difference will express the force changes before and after the participants are exposed to one of the treatments.
Time Frame: Baseline and 1 hours later (1 session of treatment), assessed as up to 1 month.
Measure: Mean (Standard Deviation); unit: Kilograms (Kg)
Arm/Group | Cathode Stimulation | Anode Stimulation | Control
Number analyzed (Participants) | 18 | 21 | 24
Kilograms (Kg) | -0.3 (5) | -0.8 (4) | -0.8 (4)

ADVERSE EVENTS:
Time Frame: Serious and/or Other (Not Including Serious) adverse events were not collected/assessed.
Description: Serious and/or Other (Not Including Serious) adverse events were not collected/assessed.
Arm/Group | Cathode Stimulation | Anode Stimulation | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No